CLINICAL TRIAL: NCT03660852
Title: Impact of a Magnetic Resonance Imaging (MRI) Scanner Exclusively Dedicated to Emergency in the Clinical Management of Patients Presenting With Diplopia or Dizziness
Acronym: IRM-DU
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7015
Record Dates: First submitted 2018-07-23; First posted 2018-09-07 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Dizziness; Diplopia; MRI; Emergency Department
MeSH Terms: conditions — Stroke; Dizziness; Diplopia; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before dedicated MRI
- After dedicated MRI

SUMMARY:
IRM-DU is a prospective observational single center study conducted in an emergency department to evaluate the impact of a MRI scanner exclusively dedicated to emergency in the clinical management of patients presenting with dizziness or diplopia.

The study will compare 2 strategies : after and before availability of a MRI scanner dedicated to emergency.

The primary endpoint is the proportion of patients with a diagnosis of stroke confirmed by imaging (MRI or Computed tomography (CT)) in the group "before implementation of the emergency MRI scanner" and the group "after implementation of the emergency MRI scanner".

The hypothesis is that the availability of a MRI scanner dedicated to emergency will improve the diagnosis of stroke in patients presenting with dizziness or diplopia, and will reduce Emergency Department stay, hospital stay and hospitalisation costs.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* non opponent to participate
* dizziness or diplopia requiring brain imaging in order to eliminate stroke

Exclusion Criteria:

* opponent to participate
* pregnant women
* recent cerebral trauma
* potentially eligible to thrombolysis
* impaired consciousness
* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
  All patients presented in ED with dizziness or diplopia are eligible to the study protocol
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Diagnosis is established on the positive signs of stroke highlighted on the CT scan or brain MRI according to the examination performed | 18 months
  Proportion of patients with a diagnosis of stroke confirmed by cerebral radiology (MRI or scan according to examination) in the pre- and post-MRI groups.

SECONDARY OUTCOMES:
Evaluate the time of care | 18 months
  Evaluate the time of care: time of realization of the examination of radiology (scanner or brain MRI), delay of passage in emergencies
Number of CT and brain MRI requested by the emergency physician in the before / after groups | 18 months
  Number of CT and brain MRI requested by the emergency physician in the before / after groups
Evaluate the usual management of vertigo and diplopia | 18 months
  Evaluate the usual management of vertigo and diplopia: number of CT and brain MRI requested by the emergency physician in the "before / after" groups; number of cerebral CT and MRI performed by the radiologist in the "before / after" groups
Evaluate the rate of new consultations in emergencies | 18 months
  Evaluate the rate of new consultations in emergencies for a neurological reason in the month following the initial care in emergencies, and the rate of new hospitalizations for the same reason
Rate of new emergency department visits for neurological | the month following initial emergency care
  Rate of new emergency department visits for neurological reasons in the month following initial emergency care
Evaluate the irradiation rate | 18 months
  Evaluate the irradiation rate related to the initial radiological examination performed during emergency care

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina GARNIER KEPKA, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kepka S, Zarca K, Lersy F, Moris M, Godet J, Deur J, Stoessel M, Muller J, Le Borgne P, Baloglu S, Fleury MC, Anheim M, Bilbault P, Bierry G, Durand Zaleski I, Kremer S. MRI dedicated to the emergency department for diplopia or dizziness: a cost-effectiveness analysis. Eur Radiol. 2022 Nov;32(11):7344-7353. doi: 10.1007/s00330-022-08791-7. Epub 2022 May 13. PMID 35554653